CLINICAL TRIAL: NCT02423850
Title: Three-dimensional Measurements for Monitoring Wound Healing of Diabetic Foot Ulcers
Brief Title: Three-dimensional Measurements of Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Line Bisgaard Jørgensen, MD, PhD student, Odense University Hospital
Other Study IDs: OUH3D02
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Foot
Keywords: Diabetic foot ulcers; Ulcer healing; Ulcer measurement; Ulcer area; Ulcer volume; 3D measurement
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetic foot ulcers: Newly referred patients with diabetic foot ulcers from the multidisciplinary clinic: University Centre for Wound healing, Odense University Hospital, Denmark.
  Interventions: Device: 3D Wound Assessment Monitor (WAM) camera

INTERVENTIONS:
Device: 3D Wound Assessment Monitor (WAM) camera — Three-dimensional wound measurement (2D area, 3D area, perimeter, volume) using 3D-WAM camera
  Other Names: 3D-WAM camera

SUMMARY:
Diabetic foot ulcers constitute an increasing health problem in Denmark concurrent with an ageing population and an increase in diabetes prevalence. Diabetic foot ulcers belong to the most serious and costly complications. Several studies have found that the size and depth of the ulcer is one of the major etiologic factors for delayed healing. Wound measurement is important in the monitoring of the wound healing process. For the last decade different 3D (three-dimensional) techniques for measuring wounds have been proposed in order to measure wound volume, but none of the technologies have been widely used. A 3D Wound Assessment Monitor (WAM) camera has been developed, which is able to measure wound size in 3D and to assess wound characteristics.

The investigators hypothesize that three-dimensional measurements of diabetic foot ulcers are feasible in the assessment of wound healing. A prospective cohort study is conducted in which newly admitted patients with a diabetic foot ulcer are included at the first visit at the multidisciplinary clinic. The patients are followed for one year or until complete wound healing, amputation or death. The four wound measurements: 2D area, 3D area, perimeter and volume are measured using the 3D-WAM camera with frequent intervals. Patient anthropometrics and wound data are collected during the study and correlated to the wound healing.

DETAILED DESCRIPTION:
Method

Newly admitted patients with a diabetic foot ulcer are included at the first visit in the multidisciplinary clinic. The data mentioned below are collected at the first visit and the following examinations are performed including 3D photos. The wound size (2D area, 3D area, perimeter and volume) are estimated from the photos using the 3D-WAM camera. The wound examination is repeated after 2, 4, 8, 12, 24, 36 and 52 weeks or until healing of the wound. The wound healing is estimated using changes in wound size per time unit. Patients are treated by standard ulcer treatment methods and are unaffected by the project per se. During the trial the different methods of treatment are noted including changes from initial treatment. The variables will be quantified after one year depending on time to heal, establishment of a chronic ulcer (non-healing after one year) or an amputation has been performed.

At baseline the following patient data will be collected:

* Demographic data: gender, age
* Smoking habits
* Time period between onset of wound to first visit in the multidisciplinary clinic
* Body Mass Index
* Comorbidity using Charlson Comorbidity Index score
* Type of diabetes, duration of diabetes
* Diabetic complications including retinopathy, albuminuria, coronary heart diseases and neuropathy

The following examinations will be performed at baseline:

* Blood pressure measurement
* Peripheral blood pressure
* Examination for neuropathy using monofilament
* Blood samples from patients with a diabetic foot ulcer

The clinical examination of the ulcer are performed at baseline and after 2, 4, 8, 12, 24, 36 and 52 weeks or until wound healing:

* Size of wound (2D area, 3D area, perimeter, volume) measured using the 3D-WAM camera
* Size of wound in 2D area using the digital imaging method with the software ImageJ
* Location of the ulcer
* Classification of ulcer: granulation, necrosis, epithelialisation
* Secretory potential
* Foot deformity
* Bone affection - if osteitis is suspected an x-ray is taken
* Signs of infection

The different types of ulcer treatment is registered for every ulcer:

* Type of bandage
* Antibiotics (local, systemic)
* Revision (method, frequency),
* Surgery

Effect variables

* Wound 2D area, 3D area, perimeter and volume
* Variation in 2D and 3D area measurements during the study period
* Percentage change in wound size after 2, 4, 8, 12, 24, 36 and 52 weeks

Endpoints

* Wound healing
* Amputations
* Chronic wound (non-healing after 1 year)
* Death

Significance

This project seeks to clarify whether 3D photos of wounds will provide accurate structural measures to illuminate the background for delayed ulcer healing, and thereby to create platform for a more evidence based treatment algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted patients with diabetic foot ulcers
* 18 years or older

Exclusion Criteria:

* Superficial wound (less than 5x5 mm with no substantial loss of subcutaneous tissue)
* Non-compliance (dementia, mental disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly admitted patients with diabetic foot ulcer to University Centre for Wound Healing, Odense University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Wound healing change quantified using the 3D-WAM camera | Photos are taken at week 0, 2, 4, 8, 12, 24, 36 and 52 weeks
  The 3D wound measurements at week 2, 4, 8, 12, 24, 36 and 52 are compared to the baseline measurement at week 0.
Wound healing change quantified using digital imaging method | Photos are taken at week 0, 2, 4, 8, 12, 24, 36 and 52 weeks
  The 2D wound measurements at week 2, 4, 8, 12, 24, 36 and 52 are compared to the baseline measurement at week 0.

SECONDARY OUTCOMES:
The variability in 2D area and 3D area measurements | Photos are taken at week 0, 2, 4, 8, 12, 24, 36 and 52 weeks
  The variability in 2D area (digital imaging method) and 3D area wound measurements (3D-WAM camera) at week 0, 2, 4, 8, 12, 24, 36 and 52 are compared
Diabetes type is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  Type 1 and 2
Diabetes duration is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  In years
BMI (kg/m2) is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  kg/m2
Charlson index score is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  In groups
HbA1c is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  mmol/mol
Ischemia is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  Ischemia is defined by ankle pressure below 70 mmHg and/or toe pressure below 45 mmHg
Neuropathy is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  Neuropathy is measured by Semmes Weinstein monofilament examination
Wound duration is compared to outcome of the wound | Baseline until healing, amputation or chronic wound (52 weeks)
  In weeks

OTHER OUTCOMES:
Quality of life (Questionaires) using 36-Item Short Form Survey (SF-36) is compared to outcome of the wound | Baseline, 24 and 52 weeks
  The higher the score the less disability

CONTACTS AND LOCATIONS:
Overall Officials: Knud Yderstræde, MD, PhD, Principal Investigator — Department of Endocrinology, Odense University Hospital
Locations (1):
- University Centre of Wound Healing, Odense University Hospital (OUH), Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided